CLINICAL TRIAL: NCT07393867
Title: Androgen-responsive POSLUMA-guided Intra-prostatic Boost (ARPEGGIO)
Brief Title: Androgen-responsive POSLUMA-guided Intra-prostatic Boost
Acronym: ARPEGGIO
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Martin T. King, MD, PhD (Other)
Collaborators: Blue Earth Diagnostics (Industry); Dana-Farber/Brigham and Women's Cancer Center (Other)
Responsible Party: Sponsor-Investigator, Martin T. King, MD, PhD, Director, Brachytherapy Clinical Operations, Associate Professor of Radiation Oncology, Harvard Medical School, Brigham and Women's Hospital
Organization: Brigham and Women's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-708
Record Dates: First submitted 2026-01-27; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Intermediate Risk Prostate Cancer; High Risk Prostate Cancer; Prostate Cancer
Keywords: POSLUMA; prostate-specific membrane antigen positron-emission tomography; PSMA-PET/CT; 18F-flotufolastat-PSMA-PET/CT scan; ADT and 18F-flotufolastat-guided focal SBRT microboost; androgen deprivation therapy and 18F-flotufolastat-guided focal SBRT microboost; neoadjuvant ADT; neoadjuvant androgen deprivation therapy; neoadjuvant ADT prior to SBRT; 18F-flotufolastat-PET/CT scans for intermediate and high risk prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Androgen Antagonists; bicalutamide; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ADT + SBRT + PSMA PET/CT Imaging (Experimental): * ADT as prescribed
  * PSMA PET/CT imaging will be completed at baseline, 8 weeks after ADT start, and at end of treatment
  * SBRT is administered starting 10 weeks after ADT start
  Interventions: Diagnostic Test: PSMA PET/CT; Drug: Androgen Deprivation Therapy (ADT) +/- bicalutamide; Radiation: Stereotactic Body Radiation Therapy (SBRT) +/- focal microboost

INTERVENTIONS:
Diagnostic Test: PSMA PET/CT — PSMA PET/CT is an imaging test that uses a radioactive tracer to highlight prostate cancer cells. Imaging will be performed at baseline, approximately eight weeks after starting ADT, and approximately 24 weeks after starting ADT (end of treatment). These scans are used to guide radiation treatment planning and assess treatment response.
Drug: Androgen Deprivation Therapy (ADT) +/- bicalutamide — ADT is used to lower testosterone levels, which can slow or shrink prostate tumors. All participants will receive approximately six months of ADT starting before radiation therapy, using injectable or oral medications. Depending on the type of ADT, participants may also receive daily bicalutamide. Bicalutamide is categorized as an antiandrogen, which means it will block the effects of testosterone and work together with ADT to slow down or shrink prostate cancer.
Radiation: Stereotactic Body Radiation Therapy (SBRT) +/- focal microboost — SBRT is a form of radiation therapy that delivers precise, high-dose radiation to the prostate over a short period of time. SBRT will be initiated 10 weeks after initiation of ADT and will be delivered in five sessions over two weeks. Based on PSMA PET/CT and MRI findings after initiation of ADT, some participants may receive an optional focal radiation microboost to areas of residual cancer. The microboost, if delivered, will be given during the same SBRT treatment sessions and will be limited by standard safety constraints.

SUMMARY:
This research study is for men with intermediate- or high-risk prostate cancer who are planning to receive hormone therapy and radiation treatment. The purpose of the study is to see whether a special type of diagnostic imaging done during hormone therapy can help doctors more accurately target remaining cancer with radiation, while avoiding areas that may no longer need extra treatment. All participants will receive standard hormone therapy and radiation therapy, along with three imaging scans, over a six-month period. The information gained from this study may help make prostate cancer radiation treatment more precise and reduce side effects for future patients.

DETAILED DESCRIPTION:
Prostate cancer is commonly treated with a combination of hormone therapy and radiation therapy. Hormone therapy, or androgen deprivation therapy (ADT), lowers testosterone levels and often shrinks or weakens prostate cancer before radiation begins. However, after hormone therapy starts, it can become harder for doctors to tell exactly where active cancer remains inside the prostate using standard imaging (typically an MRI). This study is being conducted to determine whether a newer imaging test can better identify which parts of the cancer are still active and may benefit from more focused radiation treatment.

All participants in this study will receive six months of ADT, which is part of standard care for intermediate- and high-risk prostate cancer. In addition, participants will undergo PSMA PET/CT scans, a type of imaging that highlights prostate cancer cells, as well as MRI scans. These scans will be performed at three time-points: before hormone therapy begins, approximately eight weeks after starting hormone therapy (before radiation planning), and again at 24 weeks (at the end of all treatment) to see how the cancer has responded to treatment.

Radiation therapy will begin shortly after the eight-week imaging scan. Participants will receive high-precision radiation (stereotactic body radiation therapy/SBRT) to the prostate over about two weeks. Based on the imaging results, doctors may give an extra "boost" of radiation to small areas that still show signs of active cancer. If the scans show that the cancer has responded well to hormone therapy, some patients may not need this extra boost. This approach is designed to deliver the strongest treatment where it is needed while limiting radiation to healthy tissue in order to minimize side effects.

The main goal of the study is to understand whether doctors can confidently use the mid-treatment PSMA PET/CT scan to guide radiation planning. Researchers will also monitor changes in PSA blood levels, imaging findings, treatment side effects, and patient-reported quality of life, including urinary, bowel, and sexual symptoms. Additionally, doctors participating in the study will provide feedback on how easy or difficult it is to define radiation target areas using the different scans.

Participation in this study lasts about 6 months, and all treatments provided are commonly used in prostate cancer care, with the incorporation of PSMA PET scans being the experimental component. While participants may or may not directly benefit, the results obtained from this study may help improve how radiation therapy is planned and delivered for future patients with prostate cancer, with the goal of maintaining treatment effectiveness while reducing side effects.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older.
* Eastern Oncology Group Status 0 to 1.
* Histologic diagnosis of prostate cancer.
* Prior screening MRI with at least one PI-RADS4 or PI-RADS 5 lesion, obtained within 180 days of screening.
* NCCN intermediate-risk or high-risk prostate cancer (Appendix B). All patients will be staged by MRI.
* Prior PSMA PET scan with at least one focal avid lesion greater than background prostate that is concordant with a lesion on MRI, obtained within 180 days of screening.
* Intention for SBRT (36.25 Gy/5 fraction) with focal boost (up to 50 Gy) to one MRI/PET-concordant lesion34.

Exclusion Criteria:

* Prior imaging (CT, bone scan, MRI, PSMA-PET/CT) showing nodal or distant disease.
* Intention to receive treatment intensification with secondary androgen receptor signaling inhibitors or chemotherapy.
* Clinical T4 disease.
* Prior ADT.
* Prior pelvic RT.
* Prior prostate surgery, including TURP.
* International prostate symptom score > 20.
* Prior urethral stricture.
* Prostate volume > 80 cc on MRI.
* Hip implants that cause artifacts over the prostate gland.
* Inability to discontinue anti-coagulation for fiducial marker placement.
* Active Crohn's disease or scleroderma.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with GTV treatment contours that are highly concordant with GTV-combined interim. | 8 weeks from initiation of hormone therapy/before start of radiation therapy
  To evaluate whether >50% of patients will be treated utilizing GTV contours that are highly concordant with those from interim PET/MR scans (GTV-combined-interim) based on the dice coefficient

SECONDARY OUTCOMES:
Geometric accuracies of GTV-Combined-Baseline and GTV-combined-interim contours | 8 weeks from initiation of hormone therapy/before start of radiation therapy
  The Dice coefficient of GTV-Combined-Baseline contours by the treating physician versus those independently drawn by the principal investigator will be calculated. The Dice coefficient of GTV-Combined-Interim contours by the treating physician versus those independently drawn by the principal investigator will also be calculated.
PSA response | 8 weeks from initiation of hormone therapy and 24 weeks from initiation of hormone therapy (end of treatment)
  The median PSA values at 8-weeks and 24-weeks will be evaluated. The percentage of patients with a PSA≥0.1 ng/mL will be calculated.
PSMA PET response | 8 weeks from initiation of hormone therapy and 24 weeks from initiation of hormone therapy (end of treatment)
  PSMA-PET/CT response at 8-weeks and 24-weeks will be characterized utilizing PSMA PET RECIP 1.0 criteria.
  * Complete response: Absence of any PSMA uptake at interim PET.
  * Partial: 30% or greater decrease in PSMA-avid total tumor volume.
  * Progression: 20% or greater increase in total tumor volume. New PSMA-avid lesions will also count as progression.
  * Stable disease: Less than 30% decrease or less than 20% increase in total tumor volume.
MRI ADC contrast ratio | 8 weeks from initiation of hormone therapy
  The ADC contrast ratio at baseline and 8-weeks will be calculated by evaluating the ratio of the mean ADC contrast within GTV-MRI against ADC contrast within a surrounding 2 mm ring.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at Milford Regional Medical Center, Milford, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center in Clinical Affiliation with South Shore Hospital, Weymouth, Massachusetts